CLINICAL TRIAL: NCT07373457
Title: A Single-Center, Randomized, Double-blind, Placebo-controlled, Single and Multiple Dosing, Dose-escalation, Phase 1 Clinical Trial to Evaluate the Safety, Tolerability, PK/PD, Food Effect of HW201877 in Healthy Volunteers.
Brief Title: A Phase I Study of HW201877 in Healthy Subjects
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Wuhan Humanwell Innovative Drug Research and Development Center Limited Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RFIB-I-202501
Record Dates: First submitted 2026-01-06; First posted 2026-01-28 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Healthy Participants; IBD (Inflammatory Bowel Disease)
MeSH Terms: conditions — Inflammatory Bowel Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HW201877 capsules (Experimental): Single or multiple oral doses of HW201877 capsules, and food effect of HW201877 capsules
  Interventions: Drug: HW201877 capsules
- Placebo (Placebo Comparator): Single or multiple oral doses of placebo, and food effect of placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: HW201877 capsules — Dose 1 to Dose 7
  Arms: HW201877 capsules
Drug: Placebo — Dose 1 to Dose 7
  Arms: Placebo

SUMMARY:
This is a Phase I, randomized, double-blind, placebo-controlled study to assess the safety, tolerability, pharmacokinetic (PK), pharmacodynamic (PD), and food effect (FE) of HW201877 in healthy subjects following (1) a single ascending dose (Part 1), which includes a single-dose, two-period crossover FE cohort; (2) a multiple ascending dose (Part 2).

ELIGIBILITY:
Key Inclusion Criteria:

* Before enrollment in the study, each subject shall sign the informed consent form and be fully apprised of the study content, implementation procedures and potential adverse reactions.
* Subjects are willing to voluntarily use effectivecontraceptives from screening to at least 6 months after the last dose administration.
* 18 years to 55 years (inclusive), male and female.
* Male subjects weight ≥50 kg and female subjects weight ≥45 kg. Bodymass index (BMI) : 18-28 kg/m2 (inclusive) .

Key Exclusion Criteria:

* Smoking more than 5 cigarettes per day within 3 months prior to screening.
* Allergic diathesis (with a history of allergies to multiple drugs and foods).
* A history of drug abuse and/or alcoholism (consuming 14 units of alcohol per week; 1 unit = 285 mL of beer, 25 mL of distilled spirits, or 100 mL of wine).
* Have taken any medications that alter hepatic enzyme activity within 28 days prior to screening.
* Have consumed special diets (including pitaya, mango, lime, grapefruit, carambola, orange, grapefruit or grapefruit-containing products, etc.) or engaged in strenuous exercise within 2 weeks prior to screening, or having other factors that may affect the absorption, distribution, metabolism and excretion of the study drug.
* Have taken any investigational drugs or participated in any other clinical drug trials within 3 months prior to the first administration of the study drug.
* Clinically significant abnormalities in clinical laboratory tests, or a history of clinically significant findings of the following diseases within 12 months prior to screening (including but not limited to gastrointestinal, renal, hepatic, neurological, hematological, endocrine, oncological, pulmonary, immunological, psychiatric, or cardio-cerebrovascular diseases).
* Unable to tolerate venipuncture, or with a history of needle phobia or hematophobia.
* Not suitable for this study as judged by the investigator.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 104 (Estimated)
Dates: Start 2025-06-26 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
The number and severity of treatment emergent adverse events (TEAEs) | Day 1 to Day 5
  To assess the safety and tolerability of single or multiple oral dose of HW201877 in healthy adult volunteers

CONTACTS AND LOCATIONS:
Locations (1):
- The First Hospital of Jilin University, Changchun, China

IPD SHARING:
Plan to Share IPD: No